CLINICAL TRIAL: NCT00006235
Title: A Phase I Trial of Combination Carboplatin and Lipsomal Doxorubicin (Doxil) In Recurrent Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Brief Title: Liposomal Doxorubicin and Carboplatin in Treating Patients With Recurrent Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000068160; GOG-9909
Record Dates: First submitted 2000-09-11; First posted 2004-06-22 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2006-02

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; fallopian tube cancer; primary peritoneal cavity cancer; Brenner tumor
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Carboplatin

INTERVENTIONS:
Drug: carboplatin
Drug: pegylated liposomal doxorubicin hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining liposomal doxorubicin and carboplatin in treating patients who have recurrent ovarian, fallopian tube, or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of doxorubicin HCl liposome (Doxil) when combined with carboplatin in patients with recurrent ovarian, fallopian tube, or primary peritoneal cancer. II. Determine the toxicity of this regimen in these patients. III. Determine the rate of response in patients treated with this regimen.

OUTLINE: This is a dose escalation, multicenter study of doxorubicin HCl liposome (Doxil). Patients receive Doxil IV over 1 hour and carboplatin IV on day 1. Treatment continues every 4 weeks for a minimum of 6 courses in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of Doxil until the maximum tolerated dose (MTD) is determined. The MTD is defined as the highest dose at which 0 or 1 of 6 patients experience dose limiting toxicity. Patients are followed every 3 months for 2 years, then every 6 months for 3 years, and then annually thereafter until recurrence or death.

PROJECTED ACCRUAL: Approximately 24 patients will be accrued for this study over 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven recurrent ovarian, tubal, or peritoneal cancer that is platinum sensitive (i.e., 6 months from last chemotherapy) Maximum of 1 prior chemotherapy regimen comprised of no more than 6 treatments at first recurrence Must have 1 of the following epithelial subtypes: Serous adenocarcinoma Endometrioid adenocarcinoma Mucinous adenocarcinoma Undifferentiated carcinoma Clear cell adenocarcinoma Mixed epithelial carcinoma Transitional cell Malignant Brenner tumor Adenocarcinoma not otherwise specified Measurable or evaluable disease Greater than 2 cm by CT scan, if measurable

PATIENT CHARACTERISTICS: Age: Not specified Performance status: GOG 0-2 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1,500/mm3 Hepatic: Bilirubin normal SGOT, SGPT, GGT, and alkaline phosphatase no greater than 2.5 times upper limit of normal No acute hepatitis Renal: Creatinine clearance greater than 50 mL/min Cardiovascular: LVEF normal by MUGA No congestive heart failure No unstable angina No myocardial infarction within the past 6 months Abnormal cardiac conduction (e.g., bundle branch block, heart block) allowed if disease has been stable for at least 6 months Other: No septicemia or significant infection No severe gastrointestinal bleeding No other malignancy within the past 5 years except nonmelanomatous skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior anthracycline therapy At least 3 weeks since other prior chemotherapy for ovarian, fallopian tube, or peritoneal cancer and recovered Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: At least 3 weeks since prior surgery for ovarian, fallopian tube, or peritoneal cancer and recovered Other: No other prior cancer therapy that would preclude study therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Primary Completion 2006-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rodriguez, MD, Study Chair — University Hospitals Seidman Cancer Center